CLINICAL TRIAL: NCT03459404
Title: Single-institution Case-series Analysis on the Addition of the Sufentanil NanoTab PCA System/15 mcg (Zalviso™) to a Multimodal Analgesic Regimen in Vertebral Surgery: A Preliminary Investigation
Brief Title: Sufentanil NanoTab PCA System/15 mcg for Acute Post-Operative Pain in Vertebral Surgery: A Preliminary Investigation
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, VERGARI ALESSANDRO, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: ZLV022018
Record Dates: First submitted 2018-02-20; First posted 2018-03-08 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Pain; Spinal Fusion; Spondylolisthesis, Lumbar Region; Sufentanil
MeSH Terms: conditions — Pain, Postoperative; Spondylolisthesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sufentanil NanoTab PCA System/15 mcg: Drug: Sufentanil 15 mcg
  Unless contraindicated patients also received around the clock regimen of NSAIDS (ketoprofen 200 mg/day) and acetaminophen (1000 mg every 8 hours).
  Interventions: Combination Product: Sufentanil NanoTab PCA System

INTERVENTIONS:
Combination Product: Sufentanil NanoTab PCA System — 15 mcg Sufentanil NanoTab self-administered sublingually up to every 20 minutes as needed for pain for at least 48 hours and up to 72 hours

SUMMARY:
The Zalviso® Sufentanil Sublingual Tablet System (SSTS) (Grünenthal Italia, Milan, Italy) is a patient-controlled analgesia (PCA) system approved in September 2015 by the European Commission for the management of acute moderate-to-severe pain in adult patients in a hospital setting. This preprogrammed drug/device combination product delivers a fixed dose of 15 mcg of sufentanil tablets as needed, in a non-invasive sublingual dosage form.

Multimodal analgesia is defined as the administration, by one or more routes, of various analgesic medications with different mechanisms of action, thereby providing superior analgesia with fewer side effects. To improve pain control and patient satisfaction, patient-controlled analgesia (PCA) techniques have been developed, i.e. any delivery system which allows patients to self administer predetermined doses of analgesic drug to relieve pain. Over the past decades, intravenous (IV) PCA with morphine has been the gold standard for acute pain control. In our clinical practice, though, not only IV-PCA pumps were frequently prone to technical problems, but also patients and caregivers were not often able to understand or activate them, thus raising important safety issues and profoundly affecting the management of pain control. As a consequence, IV-PCA eventually fell into disuse, although no alternative has emerged until recently. The SSTS should go beyond the above-quoted limitations: it is a non invasive, patient-controlled and easy to use device, with an effective and safe opioid profile. It is, in our thinking, a promising technology.

The aim of this retrospective analysis is to examine the role of the SSTS for management of pain after vertebral surgery, as part of a multimodal approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent elective open lumbar arthrodesis surgery (either by an anterior or posterior approach) in degenerative lumbar spine conditions who were between 18 and 75 years old and post-operatively treated with Sufentanil NanoTab PCA system as part of a multimodal analgesic regimen.
* General anesthesia was performed. Perioperative regional anesthetic techniques and local anesthetic wound infiltration in the operating room were not performed.

Exclusion criteria:

* Patients who refused to participate in the study.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who met the inclusion criteria and were operated in Policlinico A. Gemelli from September 2017 to February 2018.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Postoperative pain intensity assessed at 24 hours | NRS-11 is assessed at 24 hours.
  Pain intensity is assessed using an 11-point Numeric Rating Scale (NRS-11). It ranges from '0' representing 'no pain' to '10' representing 'the worst pain imaginable'.

SECONDARY OUTCOMES:
Postoperative pain intensity assessed at 48 hours | NRS-11 is assessed at 48 hours.
  Pain intensity is assessed using an 11-point Numeric Rating Scale (NRS-11). It ranges from '0' representing 'no pain' to '10' representing 'the worst pain imaginable'.
Patient satisfaction | At discharge (at least 48 hours)
  Satisfaction with level of pain control and satisfaction with method of administration of pain medication are scored on a 4-point scale (extremely dissatisfied to extremely satisfied).
Side effects | During the period of SSTS administration (up to 72 hours)
  Nausea, vomiting, sleepiness, itching, dizziness, others
Length of hospital stay after surgery | At least 48 hours
  Variable, depending on clinical case
Postoperative pain intensity assessed at 72 hours | NRS-11 is assessed at 72 hours.
  Pain intensity is assessed using an 11-point Numeric Rating Scale (NRS-11). It ranges from '0' representing 'no pain' to '10' representing 'the worst pain imaginable'.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Vergari, Principal Investigator — Department of Anesthesiology and Intensive Care Medicine, Fondazione Policlinico A. Gemelli, Rome
Locations (1):
- Policlinico A. Gemelli, Rome, Italy